CLINICAL TRIAL: NCT02400983
Title: Registry on Automatic Algorhitm on Atrial Capture: REAL ACap Registry
Brief Title: Real Life Automatic Atrial Capture Device Control
Status: Completed | Type: Observational
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Dr.Massimo Giammaria, MD, Maria Vittoria Hospital
Other Study IDs: 01
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Sinus Bradycardia; Sinus Node Disease; Atrio-ventricular Block; Heart Failure
Keywords: ACAP, Automatic Algorithm
MeSH Terms: conditions — Sick Sinus Syndrome; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pacemaker, ICD

SUMMARY:
The main objective of this study is to verify the effectiveness of the new ACAP ® Confirm algorithm in the automatic management of atrial capture.

ELIGIBILITY:
Inclusion Criteria:

* Patients had undergone first implantation or device replacement with a Medical device (PM, ICD, CRT-P, CRT-D) endowed with ACAP Confirm ® algorithm features between May 2011 and March 2012

Exclusion Criteria:

* Atrial fibrillation

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients had undergone first implantation or device replacement with a device (PM, ICD, CRT-P, CRT-D) endowed with ACAP Confirm ® algorithm features between May 2011 and March 2012
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The main objective of this study is to verify the effectiveness of the new ACAP Confirm ® algorithm in management of atrial capture in both new implants and patients undergoing device replacements with different manufactures atrial leads. | 6 Months

SECONDARY OUTCOMES:
Relationship with pulse width | 6 Months
Clinical equivalence of automatic and manual thresholds tests results. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Giammaria, Principal Investigator — Maria Vittoria Hospital